CLINICAL TRIAL: NCT04548986
Title: Single-center Prospective Study to Validate the Performance of the Aktiia Optical Blood Pressure Monitoring (OBPM) Device at the Wrist Against Ambulatory Blood Pressure Monitoring (ABPM)
Acronym: OBPM_ABPM2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyril Pellaton (Other)
Collaborators: Aktiia SA (Industry)
Responsible Party: Sponsor-Investigator, Cyril Pellaton, Cyril Pellaton, Hopital Neuchatelois
Organization: Hopital Neuchatelois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OBPM_ABPM2020
Record Dates: First submitted 2020-08-26; First posted 2020-09-16 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): single arm study
  Interventions: Device: Aktiia.product

INTERVENTIONS:
Device: Aktiia.product — The participants wear Aktiia.bracelet for the duration of the cardiac rehabilitation program. The device is initialized once per week.

SUMMARY:
This study aims to assess the performances of optical blood pressure monitoring device, Aktiia.product in the context of cardiac rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (aged between 21 and 65)
* Subjects fluent in written and spoken French
* Subjects enrolled in a 12-weeks cardiac rehabilitation program
* Subjects agreeing to participate
* Subjects that have signed the informed consent form

Exclusion Criteria:

* Subjects with tachycardia (heart rate at rest > 120bpm)
* Subjects with atrial fibrillation
* Subjects with severe heart failure (LVEF<35%)
* Subjects with severe renal dysfunctions (eGFR < 30mL/min/1.73 m2)
* Subjects with pheochromocytoma
* Subjects with Raynaud's disease
* Subjects with trembling and shivering
* Subjects with interarm systolic difference > 15 mmHg
* Subjects with interarm diastolic difference > 10 mmHg
* Subjects with arm paralysis
* Women in known pregnancy
* Subjects with an arteriovenous fistula
* Subjects with arm amputations
* Subjects with the upper arm circumference > 64 cm
* Subjects with the wrist circumference > 22 cm
* Subjects with the exfoliative skin diseases
* Subjects with lymphoedema

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Mean absolute error for blood pressure | up to 24 hours
  The mean absolute error between the Reference (standard ambulatory blood pressure monitor) and Aktiia.product for systolic (SYS) and diastolic (DIA) blood pressure in mmHg
Mean error for blood pressure | up to 24 hours
  The mean error between the Reference and Aktiia.product for SYS and DIA in mmHg
Standard deviation of the error for blood pressure | up to 24 hours
  The standard deviation of the error between Reference and Aktiia.product for SYS and DIA in mmHg
Mean absolute error for heart rate | up to 24 hours
  The mean absolute error between the Reference (standard ambulatory blood pressure monitor) and Aktiia.product for heart rate in bpm
Mean error for heart rate | up to 24 hours
  The mean error between the Reference and Aktiia.product for heart rate in bpm
Standard deviation of the error for heart rate | up to 24 hours
  The standard deviation of the error between Reference and Aktiia.product for heart rate in bpm

SECONDARY OUTCOMES:
Evaluation of the impact of ABPM induced stress on BP readings using inferential statistics. | 1 week
  Aktiia values acquired during the first day (with ABPM) will be compared to values acquired during other days of the week and a t-test will be performed. The analysis will be repeated for night values.
Evaluation of patient's satisfaction for the two devices through a survey with multiple questions | up to 24 hours
  10-points likert scale survey, an agree-disagree scale with minimum 0 and maximum 10. Minimum value means strong disagreement, maximum value means strong agreement.
Assessment of the calibration stability of Aktiia OBPM algorithms | 12 weeks
  Use different calibration points going from 1 to 12 weeks
Assessment of systolic and diastolic blood pressure control during a 12 weeks cardiac rehabilitation program | 12 weeks
  comparison of blood pressure determinations taken at the beginning and at the end of the program in ambulatory settings

CONTACTS AND LOCATIONS:
Locations (1):
- Réseau Hospitalier Neuchâtelois, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almeida TP, Perruchoud D, Alexandre J, Vermare P, Sola J, Shah J, Marques L, Pellaton C. Evaluation of Aktiia cuffless blood pressure monitor across 24-h, daytime, and night-time measurements versus ambulatory monitoring: a prospective, single-centre observational study. J Hypertens. 2025 Apr 1;43(4):690-697. doi: 10.1097/HJH.0000000000003960. Epub 2025 Feb 7. PMID 39927495